CLINICAL TRIAL: NCT01569958
Title: Transcranial Direct Current Stimulation as a Novel Therapeutic Approach in Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Collaborators: Catholic University, Italy (Other); Federico II University (Other); Ministero della Salute, Italy (Other)
Responsible Party: Principal Investigator, Alessandra Lugaresi, Prof, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDCS2011-01; RF-ABR-2007-631680 (Other Grant/Funding Number: Italian Ministry of Health/RF-ABR-2007-631680)
Record Dates: First submitted 2012-03-09; First posted 2012-04-03 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tDCS (Active Comparator)
  Interventions: Other: transcranial direct current stimulation
- sham (Sham Comparator)
  Interventions: Other: Sham stimulation

INTERVENTIONS:
Other: transcranial direct current stimulation — transcranial direct current stimulation applied to the motor cortex of both sides (1 mA, 20 minutes) for five consecutive days every month for 12 months
  Arms: tDCS
Other: Sham stimulation — 1 mA stimulation for 30 seconds every 900 seconds per session
  Arms: sham

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a neurodegenerative disease characterized by progressive weakness and muscular atrophy due to the degeneration and loss of motor neurons, the nerve cells that, in the central nervous system (motor cortex, brainstem and spinal chord), control voluntary movement. Riluzole, the only drug approved for ALS treatment, modestly slow disease progression.

Transcranial direct current stimulation (tDCS) is a noninvasive technique of neuromodulation that is currently studied as a possible therapeutic tool for several neurological and psychiatric diseases and has been found safe and well tolerated. Based on experimental evidence in animals and human subjects, tDCS is expected to reduce motor cortex excitability and excitotoxicity, that is neuronal injury induced by excessive glutamatergic stimulation, one of postulated pathophysiological mechanisms in ALS.

This study will investigate if transcranial direct current stimulation of motor cortex is useful in delaying disease progression and is well tolerated in ALS patients.

DETAILED DESCRIPTION:
This is a double blind, randomized, placebo-controlled clinical trial.

Cathodic tDCS (1 mA for 20 minutes) will be sequentially applied over the motor cortex of both sides, for five consecutive days every month for twelve months. The control group will receive a sham stimulation that reproduce tactile sensation of real stimulation but has no effects on central nervous system. For stimulation, researchers will employ a CE-certified medical device acting as a micro-processor-controlled constant current source. All patients will take riluzole during the entire period of the study.

Fifty-four participants will be recruited from three Italian Centers and randomized to one of two arms of the study.

Disease progression and quality of life will be evaluated at baseline and every three months during the study.

At each visit adverse events will be reported and tolerability will be assessed through a specific questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of probable, laboratory-supported probable, or definite amyotrophic lateral sclerosis according to the El Escorial revised criteria
* spinal onset
* aged 18 to 85 years inclusive
* disease duration ≤ 24 months
* disease progression in the past 3 months
* FVC ≥ 70% of predicted
* score ≥ 2 at the item "swallowing"of the ALS Functional Rating Scale Revised
* score ≥ 2 at the item "walking"of the ALS Functional Rating Scale Revised
* in treatment with steady regimen of riluzole for a minimum of 1 month before study entry, and desiring its continuation
* able to give informed consent
* written informed consent

Exclusion Criteria:

* bulbar onset
* previous poliomyelitis
* motor neuron diseases other than ALS
* clinical involvement of other neurological systems
* pregnancy, lactation,or unwillingness to contraception if required
* possible contraindications to tDCS: metals in the head (excluding the mouth); electromedical devices; seizures; drugs or neurological conditions lowering seizure threshold; alcoholism; severe heart diseases
* any severe disease other than ALS
* experimental drugs within 1 month prior to enrollment
* drugs potentially modifying the response to tDCS

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Decline of ALSFRS-R (ALS functional rating scale-revised) from baseline to 12 months | 12 months

SECONDARY OUTCOMES:
Decline of muscle strength from baseline to 12 months | 12 months
  A megascore will be obtained by summing scores of single muscles manually tested according to the Medical Research Council Scale
Change of upper motor neuron signs from baseline to 12 months | 12 months
  A score will be obtained based on presence/absence of listed upper motor neuron signs and grade of spasticity
Decline of forced vital capacity (percent of predicted normal) from baseline to 12 months | 12 months
Change of quality of life from baseline to 12 months | 12 months
  The ALSAQ-40 questionnaire will be employed

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Lugaresi, MD, PhD, Principal Investigator — Università "G. d'Annunzio" di Chieti e Pescara, Dipartimento Neuroscienze ed Imaging, and ASL n. 2 Lanciano-Vasto-Chieti
Locations (3):
- Italy (3):
  - Centro Regionale Malattie Neuromuscolari, Ospedale Clinicizzato "SS. Annunziata", Chieti, Chieti
  - Azienda Policlinico Università Federico II, Napoli, Napoli
  - Policlinico Universitario Agostino Gemelli, Rome, Rome